CLINICAL TRIAL: NCT02729454
Title: Effects of Mental Practice on the March and the Risk of Falls in People With Parkinson's Disease
Brief Title: Mental Practice in Parkinson's Disease
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Universidade Federal de Pernambuco (Other)
Responsible Party: Principal Investigator, LILIANE PEREIRA DA SILVA, Principal Investigator, Universidade Federal de Pernambuco
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: CAAE 46155315.3.0000.5208
Record Dates: First submitted 2016-03-26; First posted 2016-04-06 (Estimated); Last update posted 2016-09-28 (Estimated); Status verified 2016-09

CONDITIONS: Parkinson Disease
MeSH Terms: conditions — Parkinson Disease | interventions — Physical Therapy Modalities

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Exclusively physical therapy (Active Comparator): The patients will be submitted to 15 therapeutical sessions two times per week with length of 40 minutes for motor physiotherapy . Each session of the motor physiotherapy will be constituted of exercises that include stretching (emphasizing the front of the torso), reinforcement (with emphasis in inferior members extensores); active exercises as transference (for example, to put into motion it bed or uprising of a chair), to reach and to grasp and training of balance and march.
  Interventions: Other: physical therapy
- Mental Practice And Physical Therapy (Experimental): In the group submitted to the mental Practice the sessions will be individualized and occur in tranquil room after physical therapy (Same performed with the control group). During the mental practice the patient will be guided to stand, where he will be requested initially to identify and to sequencer the necessary joints for the accomplishment of an only step, being they:flexion of the thigh and leg rights, extension of the right leg more dorsiflexed of the right foot; touch of the heel and discharge of weight of the right foot and inclined body to the front. The sessions occur two times per week during 15 minutes.
  Interventions: Other: Mental practice and physical therapy

INTERVENTIONS:
Other: Mental practice and physical therapy
  Arms: Mental Practice And Physical Therapy
Other: physical therapy
  Arms: Exclusively physical therapy

SUMMARY:
Introduction Although drug therapy is the mainstay of treatment for Parkinson's disease, the therapy also has its importance by means of exercises which maintains the muscular activity and preserve mobility. One of the techniques that has been used for physical therapy is the mental practice of the mental simulation of movement, aiming at learning or improvement of motor skills through the cortex areas of activation responsible for the movement of preparation before it is executed. In patients with Parkinson's disease motor anticipation this system is compromised, culminating in the march changes and increased risk of falls. Objective: To evaluate the effects of mental practice on physical therapy on the march and the risk of falls in people with Parkinson's disease. Method: The study is defined as a randomized clinical trial with systematic recruitment. Recruitment will be conducted at the Clinic of Neurology, Hospital das clinics Federal University of Pernambuco (Pro-Parkinson Project: Neurology) and the intervention will be held at the same hospital physiotherapy clinic. Both the control group and the trial will be subjected to 15 therapy sessions twice a week, lasting 40 minutes for physical therapy and 15 for mental practice.

ELIGIBILITY:
Inclusion Criteria:

* Patients with clinical diagnosis of idiopathic Parkinson's disease
* Male and female
* Stage 1-3 of the Hoehn and Yahr scale.

Exclusion Criteria:

* Have other neurological diseases
* They have decompensated systemic diseases
* Musculoskeletal changes that prevent the achievement of movements
* With lowering of the cognitive level assessed using the Mini-Mental State Examination with cutoff point according to education
* With respiratory impairment
* With medical restrictions for performing exercises
* Do not get hold motor imagination during the application of Visual and Kinesthetic Imagery Questionnaire-10
* In physical therapy, occupational therapy service for 3 months or more;
* Patients with moderate to severe depression assessed by inventory Beck Depression Inventory

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 18 (Actual)
Dates: Start 2015-10; Primary Completion 2016-09 (Actual); Study Completion 2016-09 (Actual)

PRIMARY OUTCOMES:
Dynamic Gait Index test to evaluate gait and risk of falls | two months
  It is an instrument of functional mobility assessment, the Dynamic Gait Index (DGI), aims to evaluate and document the patient's ability to modify the march in response to changing demands of certain tasks. DGI consists of eight tasks involving gait in different sensorial contexts, which include flat surface, changes in gait speed, horizontal and vertical movements of the head, go over and around obstacles; turn on your own body axis, up and down stairs. Each patients is assessed by means of an ordinal scale with 4 categories and scored according to his/her own performance in each task: 3 = normal gait, 2 = slight impairment, 1 = moderate impairment and 0 = severe impairment. Maximum scoring is 24 points, and a score of 19 points or less is able to predict a risk of falls.
  Praz
Timed up and go Test to evaluate risk of falls | two months
  The Tine up and Go Test (TUG) is used to assess risk of falls. To perform the test the patient will be instructed to sit with his back on an unsupported chair arms and the examiner will give the verbal command "go" in which the patient will get up and go a distance of three meters , returning and sitting in the same chair with your back supported.Shorter values than 10 seconds to perform the test indicate low risk of falls, values between 10 to 20 seconds indicate medium risk of falls and greater than 20 seconds represent high risk for falls
Walk Test of 10 meters to evaluate gait | two months
  The walk test of 10 m is a tool used to evaluate the spatial and temporal attributes kinematic gait, as it will be evaluated the average speed of travel, number of steps and cadence. For the test will be placed markers in position 2 and 8 m. The patient will be instructed to walk at a comfortable pace from one extreme to another. A physical therapist will use the stopwatch to determine how long it takes for the patient to go through the central 6 meters of the route.
history questionnaire falls to evaluate risk of falls | two months
  The falls of history questionnaire seeks reports of falls occurred in the patient's daily life and contains the following questions: 1. Have you fallen or stumbled in the last 12 months, for any reason, even if it is not related to Parkinson's disease? 2. How many times have you fallen in the last 12 months (daily / weekly / monthly / etc)? 3. Are you afraid of falling? If dropped, question to clarify, for each fall (or default): 4. Where were you when he fell? 5. What were you doing or trying to do at the moment? 6. What do you think caused the fall? 7. Did you lose consciousness before the fall? 8. What pattern can be identified in the fall? 9. You showed balance and nearly fell last year? 10. How often have you had balance and nearly fell last year? In case of almost fall, are asked to clarify the pattern: 11. What kinds of things do you usually do when out of balance and almost fall? 12. Why do you think that you almost fall? 13. How do you avoid the drop this time?

CONTACTS AND LOCATIONS:
Locations (1):
- Hospital Das Clinicas - Ufpe, Recife, Pernambuco, Brazil

IPD SHARING:
Plan to Share IPD: No